CLINICAL TRIAL: NCT01988935
Title: Integrated PTSD and Smoking Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mark B. Powers, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K01DA035930 (NIH); NCT01857739 (obsolete NCT alias)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged Exposure + Smoking Cessation (Experimental): Prolonged Exposure therapy plus smoking cessation intervention
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Smoking Cessation
- Smoking Cessation (Active Comparator): Smoking cessation intervention
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Prolonged Exposure — Weekly psychotherapy sessions x 12 weeks, focused on gradually confronting distressing trauma-related memories and reminders.
  Arms: Prolonged Exposure + Smoking Cessation
Behavioral: Smoking Cessation — Weekly smoking cessation counseling (cognitive behavioral therapy) plus the nicotine patch to reduce withdrawal symptoms.

SUMMARY:
Research shows that people with PTSD are more likely to smoke than people without PTSD. It also shows that people with PTSD have more difficulty at attempts to quit smoking. This study is part of a program aimed at finding out how best to help smokers quit who also have PTSD. One option is to give patients standard smoking cessation treatment including nicotine replacement and cognitive behavioral therapy. Another option is to give patients the standard smoking cessation treatment in addition to treatment for their PTSD symptoms (called prolonged exposure). However, it is not known which method works better. In order to answer this question, patients will be assigned by chance to one of two groups. One group will be given standard smoking cessation treatment to help quit smoking. A second group will be given the standard smoking cessation intervention to help quit smoking in addition to a form of psychotherapy called Prolonged Exposure to reduce symptoms of PTSD. The patients will be randomly assigned (by chance) to one of these groups. If the patient is assigned to the smoking cessation only condition and the patient still has PTSD symptoms after the last study visit (week 30) the patient will be offered treatment for your PTSD symptoms (Prolonged Exposure) at no cost. The patient's participation will help the investigators determine if treating PTSD symptoms enhances the ability of standard smoking cessation to help people quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* You have PTSD
* You currently smoke more than 8 cigarettes per day
* You have a motivation to quit smoking
* You are between the age of 18 and 65.

Exclusion Criteria:

* You are currently using other tobacco products (other than cigarettes)
* You have any history of a suicide attempt, or are at significant risk of self-harm or harm to others
* You have severe depression
* You have any history of bipolar disorder, psychotic disorder
* You have a diagnosis of eating disorder, or substance abuse or dependence (excluding nicotine) within the past six months
* You are currently receiving other treatment specifically for PTSD or smoking cessation
* You are unable to read and speak English (as the materials are provided in English)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Smoking Status | 3 months

SECONDARY OUTCOMES:
PTSD Symptoms | 3 months
General Mood and Anxiety Symptoms | 3 months
Side Effects | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States